CLINICAL TRIAL: NCT02163447
Title: Reducing the Burden of Malaria in HIV-uninfected Pregnant Women and Infants (PROMOTE Birth Cohort 1)
Brief Title: Reducing the Burden of Malaria in HIV-uninfected Pregnant Women and Infants
Acronym: PROMOTE-BC1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Grant Dorsey, M.D, Ph.D. (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor-Investigator, Grant Dorsey, M.D, Ph.D., Professor, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PROMOTE-BC1; P01HD059454 (NIH)
Record Dates: First submitted 2014-06-05; First posted 2014-06-13 (Estimated); Results first posted 2018-11-14 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Malaria
Keywords: Chemoprevention; Malaria; Uganda; Sulfadoxine-pyrimethamine; Dihydroartemisinin-piperaquine
MeSH Terms: conditions — Malaria | interventions — fanasil, pyrimethamine drug combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- 3 dose SP pregnancy / 3 monthly DP infancy (Active Comparator): Women will be given SP (3 full strength tabs, 500 mg/25 mg) 3 times during pregnancy at 20, 28, and 36 weeks gestational age. In addition, placebos will be used to mimic the identical dosing strategy such that every 4 weeks women will receive two pills on day 1 (SP and placebo, DP and placebo, or two placebos) followed by one pill on days 2 and 3 (DP or placebo). Two placebos will be used, one that mimics the appearance of SP and one that mimics the appearance of DP.
  Infants will be given DP (once a day for 3 consecutive days using weight-based guidelines) every 12 weeks between 8 and 104 weeks of age. Infants randomized to receive DP every 12 weeks will receive placebo mimicking the dosing of DP every 4 weeks when they are not receiving study drug.
  Interventions: Drug: 3 dose sulfadoxine-pyrimethamine (SP) for adult women during pregnancy; Drug: 3-monthly dihydroartemisinin-piperaquine (DP) for infants
- 3 dose DP pregnancy / 3 monthly DP infancy (Active Comparator): Women will be given DP (3 full strength tabs, 40 mg/320 mg, given once a day for 3 consecutive days) 3 times during pregnancy at 20, 28, and 36 weeks gestational age. In addition, placebos will be used to mimic the identical dosing strategy such that every 4 weeks women will receive two pills on day 1 (SP and placebo, DP and placebo, or two placebos) followed by one pill on days 2 and 3 (DP or placebo). Two placebos will be used, one that mimics the appearance of SP and one that mimics the appearance of DP.
  Infants will be given DP (once a day for 3 consecutive days using weight-based guidelines) every 12 weeks between 8 and 104 weeks of age. Infants randomized to receive DP every 12 weeks will receive placebo mimicking the dosing of DP every 4 weeks when they are not receiving study drug.
  Interventions: Drug: 3 dose dihydroartemisinin-piperaquine (DP) for adult women during pregnancy; Drug: 3-monthly dihydroartemisinin-piperaquine (DP) for infants
- 3 dose DP pregnancy / monthly DP infancy (Active Comparator): Women will be given DP (3 full strength tabs, 40 mg/320 mg, given once a day for 3 consecutive days) 3 times during pregnancy at 20, 28, and 36 weeks gestational age. In addition, placebos will be used to mimic the identical dosing strategy such that every 4 weeks women will receive two pills on day 1 (SP and placebo, DP and placebo, or two placebos) followed by one pill on days 2 and 3 (DP or placebo). Two placebos will be used, one that mimics the appearance of SP and one that mimics the appearance of DP.
  Infants will be given DP (once a day for 3 consecutive days using weight-based guidelines) every 4 weeks between 8 and 104 weeks of age.
  Interventions: Drug: 3 dose dihydroartemisinin-piperaquine (DP) for adult women during pregnancy; Drug: Monthly dihydroartemisinin-piperaquine (DP) for infants
- monthly DP pregnancy / 3 monthly DP infancy (Active Comparator): Women will be given DP (3 full strength tabs, 40 mg/320 mg, given once a day for 3 consecutive days) every 4 weeks during pregnancy. In addition, placebos will be used to mimic the identical dosing strategy such that every 4 weeks women will receive two pills on day 1 (SP and placebo, DP and placebo, or two placebos) followed by one pill on days 2 and 3 (DP or placebo). Two placebos will be used, one that mimics the appearance of SP and one that mimics the appearance of DP.
  Infants will be given DP (once a day for 3 consecutive days) every 12 weeks between 8 and 104 weeks of age. Infants randomized to receive DP every 12 weeks will receive placebo mimicking the dosing of DP every 4 weeks when they are not receiving study drug.
  Interventions: Drug: Monthly dihydroartemisinin-piperaquine (DP) for adult women during pregnancy; Drug: 3-monthly dihydroartemisinin-piperaquine (DP) for infants
- monthly DP pregnancy / monthly DP infancy (Active Comparator): Women will be given DP (3 full strength tabs, 40 mg/320 mg, given once a day for 3 consecutive days) every 4 weeks during pregnancy. In addition, placebos will be used to mimic the identical dosing strategy such that every 4 weeks women will receive two pills on day 1 (SP and placebo, DP and placebo, or two placebos) followed by one pill on days 2 and 3 (DP or placebo). Two placebos will be used, one that mimics the appearance of SP and one that mimics the appearance of DP.
  Infants will be given DP (once a day for 3 consecutive days) every 4 weeks between 8 and 104 weeks of age.
  Interventions: Drug: Monthly dihydroartemisinin-piperaquine (DP) for adult women during pregnancy; Drug: Monthly dihydroartemisinin-piperaquine (DP) for infants

INTERVENTIONS:
Drug: Monthly dihydroartemisinin-piperaquine (DP) for adult women during pregnancy
  Other Names: Duo-Cotexin (Holley-Cotec)
  Arms: monthly DP pregnancy / 3 monthly DP infancy; monthly DP pregnancy / monthly DP infancy
Drug: 3 dose dihydroartemisinin-piperaquine (DP) for adult women during pregnancy
  Other Names: Duo-Cotexin (Holley-Cotec)
  Arms: 3 dose DP pregnancy / 3 monthly DP infancy; 3 dose DP pregnancy / monthly DP infancy
Drug: 3 dose sulfadoxine-pyrimethamine (SP) for adult women during pregnancy
  Other Names: Kamsidar (KPI)
  Arms: 3 dose SP pregnancy / 3 monthly DP infancy
Drug: Monthly dihydroartemisinin-piperaquine (DP) for infants
  Other Names: Duo-Cotexin (Holley-Cotec)
  Arms: 3 dose DP pregnancy / monthly DP infancy; monthly DP pregnancy / monthly DP infancy
Drug: 3-monthly dihydroartemisinin-piperaquine (DP) for infants
  Other Names: Duo-Cotexin (Holley-Cotec)
  Arms: 3 dose DP pregnancy / 3 monthly DP infancy; 3 dose SP pregnancy / 3 monthly DP infancy; monthly DP pregnancy / 3 monthly DP infancy

SUMMARY:
This will be a double-blinded randomized controlled phase III trial of 300 HIV uninfected pregnant women and the children born to them. The study interventions will be divided into two phases. In the first phase, HIV uninfected women at 12-20 weeks gestation will be randomized in equal proportions to one of three intermittent preventive therapy in pregnancy (IPTp) treatment arms: 1) 3 doses of sulfadoxine-pyrimethamine (SP), 2) 3 doses of dihydroartemisinin-piperaquine (DP), or 3) monthly DP. All three interventions arms will have either SP or DP placebo to ensure adequate blinding is achieved. Follow-up for the pregnant women will end approximately 6 weeks after giving birth. In the second phase of the study, all children born to mothers enrolled in the study will be followed from birth until they reach 36 months of age. Children born to mothers randomized to receive 3 doses of SP during pregnancy will receive DP every 3 months between 2-24 months of age. Children born to mothers randomized to receive 3 doses of DP or monthly DP during pregnancy will receive either DP every 3 months or monthly DP between 2-24 months of age. To ensure adequate blinding, children who will receive DP every 3 months will be given DP placebo during the months they will not be taking DP. Children will then be followed an additional year between 24-36 months of age following the interventions. We will test the hypothesis that IPT with DP will significantly reduce the burden of malaria in pregnancy and infancy and improve the development of naturally acquired antimalarial immunity.

DETAILED DESCRIPTION:
Pregnant women will be scheduled to be seen in the clinic every 4 weeks during their pregnancy and 6 weeks following delivery. In addition, pregnant women will be instructed to come to the study clinic for all their medical care and avoid the use of any outside medications. Children will be scheduled to be seen in the clinic every 4 weeks and parents /guardians of children will be instructed to bring their child to the study clinic for all medical care and avoid the use of any outside medications. The study clinic will remain open 7 days a week from 8 a.m. to 5 p.m.

Each time a study participant is seen in the clinic a standardized history and physical exam will be performed. Patients who are febrile (tympanic temperature > 3 8.0˚C) or report history of fever in the past 24 hours will have blood obtained by finger prick for a thick blood smear. If the thick blood smear is positive, the patient will be diagnosed with malaria. If the thick blood smear is negative, the patient will be managed by study physicians for a non-malarial febrile illness. If the patient is afebrile and does not report a recent fever, a thick blood smear will not be obtained, except when following routine testing schedules.

Routine assessments will be done in the clinic every 4 weeks for both pregnant women and children. Pregnant women and children will receive standards of care as designated in the Uganda MOH guidelines. Routine care in children will use Integrated Management of Childhood Illness (IMCI) guidelines. During routine assessments subjects will be asked about visits to outside health facilities and the use of any medications outside the study protocol. Standardized assessment of adherence will also be done for study drugs administered at home and Insecticide Treated Net use. A routine history and physical exam will be performed using a standardized clinical assessment form. Blood will be collected by finger prick for thick smear, collection of plasma for PK studies, and filter paper samples. Phlebotomy for routine laboratory tests (CBC and ALT) to monitor for potential adverse events from study medications and for immunology studies will be performed every 8 weeks in pregnant women and every 16 weeks in children. Non malaria screening will also include stool ova and parasite examination, circulating filarial antigens (by ICT card for Wucheria), and blood smear for microfilaremia (including Mansonella perstans) using Knott's technique. For pregnant women and children 2-24 months of age, study drugs will be administered at the time of each routine visit.

ELIGIBILITY:
Inclusion Criteria:

1. Pregnancy confirmed by positive urine pregnancy test or intrauterine pregnancy by ultrasound
2. Estimated gestational age between 12-20 weeks
3. Confirmed to be HIV uninfected by rapid test
4. 16 years of age or older
5. Residency within 30km of the study clinic
6. Provision of informed consent by the pregnant woman for herself and her unborn child
7. Agreement to come to the study clinic for any febrile episode or other illness and avoid medications given outside the study protocol
8. Plan to deliver in the hospital

Exclusion Criteria:

1. History of serious adverse event to SP or DP
2. Active medical problem requiring inpatient evaluation at the time of screening
3. Intention of moving more than 30km from the study clinic
4. Chronic medical condition requiring frequent medical attention
5. Prior SP preventive therapy or any other antimalarial therapy during this pregnancy
6. Early or active labor (documented by cervical change with uterine contractions)

Min Age: 16 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2014-06-23 (Actual); Primary Completion 2018-05-14 (Actual); Study Completion 2018-05-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Grant Dorsey, MD, PhD, Principal Investigator — University of California, San Francisco; Diane V Havlir, MD, Principal Investigator — University of California, San Francisco; Moses Kamya, MBChB, MMed, PhD, Principal Investigator — Makerere University; Infectious Diseases Research Collaboration
Locations (1):
- IDRC Research Clinic -Tororo District Hospital, Tororo, Uganda

REFERENCES:
- [Result] Kakuru A, Jagannathan P, Muhindo MK, Natureeba P, Awori P, Nakalembe M, Opira B, Olwoch P, Ategeka J, Nayebare P, Clark TD, Feeney ME, Charlebois ED, Rizzuto G, Muehlenbachs A, Havlir DV, Kamya MR, Dorsey G. Dihydroartemisinin-Piperaquine for the Prevention of Malaria in Pregnancy. N Engl J Med. 2016 Mar 10;374(10):928-39. doi: 10.1056/NEJMoa1509150. PMID 26962728
- [Result] Muhindo MK, Kakuru A, Natureeba P, Awori P, Olwoch P, Ategeka J, Nayebare P, Clark TD, Muehlenbachs A, Roh M, Mpeka B, Greenhouse B, Havlir DV, Kamya MR, Dorsey G, Jagannathan P. Reductions in malaria in pregnancy and adverse birth outcomes following indoor residual spraying of insecticide in Uganda. Malar J. 2016 Aug 26;15(1):437. doi: 10.1186/s12936-016-1489-x. PMID 27566109
- [Result] Conrad MD, Mota D, Foster M, Tukwasibwe S, Legac J, Tumwebaze P, Whalen M, Kakuru A, Nayebare P, Wallender E, Havlir DV, Jagannathan P, Huang L, Aweeka F, Kamya MR, Dorsey G, Rosenthal PJ. Impact of Intermittent Preventive Treatment During Pregnancy on Plasmodium falciparum Drug Resistance-Mediating Polymorphisms in Uganda. J Infect Dis. 2017 Nov 15;216(8):1008-1017. doi: 10.1093/infdis/jix421. PMID 28968782
- [Result] Kapisi J, Kakuru A, Jagannathan P, Muhindo MK, Natureeba P, Awori P, Nakalembe M, Ssekitoleko R, Olwoch P, Ategeka J, Nayebare P, Clark TD, Rizzuto G, Muehlenbachs A, Havlir DV, Kamya MR, Dorsey G, Gaw SL. Relationships between infection with Plasmodium falciparum during pregnancy, measures of placental malaria, and adverse birth outcomes. Malar J. 2017 Oct 5;16(1):400. doi: 10.1186/s12936-017-2040-4. PMID 28982374
- [Result] Jagannathan P, Kakuru A, Okiring J, Muhindo MK, Natureeba P, Nakalembe M, Opira B, Olwoch P, Nankya F, Ssewanyana I, Tetteh K, Drakeley C, Beeson J, Reiling L, Clark TD, Rodriguez-Barraquer I, Greenhouse B, Wallender E, Aweeka F, Prahl M, Charlebois ED, Feeney ME, Havlir DV, Kamya MR, Dorsey G. Dihydroartemisinin-piperaquine for intermittent preventive treatment of malaria during pregnancy and risk of malaria in early childhood: A randomized controlled trial. PLoS Med. 2018 Jul 17;15(7):e1002606. doi: 10.1371/journal.pmed.1002606. eCollection 2018 Jul. PMID 30016328
- [Result] Muhindo MK, Jagannathan P, Kakuru A, Opira B, Olwoch P, Okiring J, Nalugo N, Clark TD, Ruel T, Charlebois E, Feeney ME, Havlir DV, Dorsey G, Kamya MR. Intermittent preventive treatment with dihydroartemisinin-piperaquine and risk of malaria following cessation in young Ugandan children: a double-blind, randomised, controlled trial. Lancet Infect Dis. 2019 Sep;19(9):962-972. doi: 10.1016/S1473-3099(19)30299-3. Epub 2019 Jul 12. PMID 31307883
- [Result] Conroy AL, Bangirana P, Muhindo MK, Kakuru A, Jagannathan P, Opoka RO, Liechty EA, Nakalembe M, Kamya MR, Dorsey G, John CC. Case Report: Birth Outcome and Neurodevelopment in Placental Malaria Discordant Twins. Am J Trop Med Hyg. 2019 Mar;100(3):552-555. doi: 10.4269/ajtmh.18-0659. PMID 30628574
- [Derived] Wallender E, Ali AM, Hughes E, Kakuru A, Jagannathan P, Muhindo MK, Opira B, Whalen M, Huang L, Duvalsaint M, Legac J, Kamya MR, Dorsey G, Aweeka F, Rosenthal PJ, Savic RM. Identifying an optimal dihydroartemisinin-piperaquine dosing regimen for malaria prevention in young Ugandan children. Nat Commun. 2021 Nov 18;12(1):6714. doi: 10.1038/s41467-021-27051-8. PMID 34795281
- [Derived] Hughes E, Imperial M, Wallender E, Kajubi R, Huang L, Jagannathan P, Zhang N, Kakuru A, Natureeba P, Mwima MW, Muhindo M, Mwebaza N, Clark TD, Opira B, Nakalembe M, Havlir D, Kamya M, Rosenthal PJ, Dorsey G, Aweeka F, Savic RM. Piperaquine Exposure Is Altered by Pregnancy, HIV, and Nutritional Status in Ugandan Women. Antimicrob Agents Chemother. 2020 Nov 17;64(12):e01013-20. doi: 10.1128/AAC.01013-20. Print 2020 Nov 17. PMID 33020153
- [Derived] Whalen ME, Kajubi R, Chamankhah N, Huang L, Orukan F, Wallender E, Kamya MR, Dorsey G, Jagannathan P, Rosenthal PJ, Mwebaza N, Aweeka FT. Reduced Exposure to Piperaquine, Compared to Adults, in Young Children Receiving Dihydroartemisinin-Piperaquine as Malaria Chemoprevention. Clin Pharmacol Ther. 2019 Dec;106(6):1310-1318. doi: 10.1002/cpt.1534. Epub 2019 Jul 22. PMID 31173649
- [Derived] Savic RM, Jagannathan P, Kajubi R, Huang L, Zhang N, Were M, Kakuru A, Muhindo MK, Mwebaza N, Wallender E, Clark TD, Opira B, Kamya M, Havlir DV, Rosenthal PJ, Dorsey G, Aweeka FT. Intermittent Preventive Treatment for Malaria in Pregnancy: Optimization of Target Concentrations of Dihydroartemisinin-Piperaquine. Clin Infect Dis. 2018 Sep 14;67(7):1079-1088. doi: 10.1093/cid/ciy218. PMID 29547881

RESULTS

PARTICIPANT FLOW:
Groups:
- Mothers - 3 Dose SP: Sulfadoxine-Pyrimethamine 500mg/25mg
- Mothers - 3 Dose DP: Dihydrioartemisinin-Piperaquine 40mg/320mg
- Mothers - Monthly DP: Dihydroartemisinin-Piperaquine 20mg/160mg
Period: Overall Study
Arm/Group | Mothers - 3 Dose SP | Mothers - 3 Dose DP | Mothers - Monthly DP
Started | 106 | 94 | 100
Infants Born | 101 | 93 | 100
Completed | 100 | 88 | 97
Not Completed | 6 | 6 | 3
Not completed — Withdrawal by Subject | 2 | 0 | 1
Not completed — Lost to Follow-up | 1 | 3 | 0
Not completed — Moved out of study area | 2 | 3 | 2
Not completed — Became HIV infected at time of delivery | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mothers - 3 Dose SP | Mothers - 3 Dose DP | Mothers - Monthly DP | Total
Number analyzed (Participants) | 106 | 94 | 100 | 300
Age, Continuous [Mean (Standard Deviation); unit: years] | 21.3 (3.6) | 22.2 (4.3) | 22.6 (4.0) | 22.0 (4.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 106 | 94 | 100 | 300
  Male | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 106 | 94 | 100 | 300
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Gestation (weeks) [Count of Participants; unit: Participants]
  12 to 16 wk | 75 | 65 | 67 | 207
  > 16 to 20 wk | 31 | 29 | 33 | 93
Gravidity [Count of Participants; unit: Participants]
  1 | 42 | 33 | 36 | 111
  2 | 32 | 28 | 28 | 88
  >= 3 | 32 | 33 | 36 | 101
Bed-net ownership [Count of Participants; unit: Participants]
  None | 13 | 8 | 9 | 30
  Untreated Net | 1 | 6 | 2 | 9
  Long lasting insecticide- treated net | 92 | 80 | 89 | 261
Household wealth index [Count of Participants; unit: Participants]
  Lowest third | 38 | 29 | 33 | 100
  Middle third | 32 | 37 | 31 | 100
  Highest third | 36 | 28 | 36 | 100
Weight (kg) [Mean (Standard Deviation); unit: kg] | 55.4 (6.8) | 55.6 (7.0) | 55.5 (7.5) | 55.5 (7.1)
Height (cm) [Mean (Standard Deviation); unit: cm] | 162.8 (6.8) | 162.5 (6.7) | 162.3 (7.7) | 162.5 (7.1)
White blood cells per mm^3 [Mean (Standard Deviation); unit: cells per mm^3] | 6036 (2070) | 6279 (1713) | 6040 (1572) | 6113 (1802)
Neutrophil cells per mm^3 [Mean (Standard Deviation); unit: cells per mm^3] | 3330 (1477) | 3558 (1304) | 3351 (1175) | 3409 (1327)
Platelet cells per mm^3 [Mean (Standard Deviation); unit: cells per mm^3] | 198906 (60665) | 201809 (67358) | 195840 (59593) | 198793 (62332)
Hemoglobin level g/dL [Mean (Standard Deviation); unit: g/DL] | 11.8 (1.5) | 11.9 (1.1) | 12.0 (1.4) | 11.9 (1.3)
Alanine aminotransferase level IU/L [Mean (Standard Deviation); unit: IU/L] | 15.4 (7.5) | 14.9 (5.8) | 14.7 (5.6) | 15.0 (6.4)
Detection of malaria parasites by LAMP [Count of Participants; unit: Participants]
  Yes | 59 | 55 | 57 | 171
  No | 47 | 38 | 43 | 128
  No sample collected | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Prevalence of Placental Malaria
Description: Prevalence of placental malaria based on placental histopathology dichotomized into any evidence of placental infection (parasites or pigment) vs. no evidence and by histopathology as a categorical variable based on Rogerson et al criteria.
Time Frame: Delivery
Population: Only women who delivered and had histopathology results were analyzed. 2 women in 3 Dose SP and 1 woman in monthly DP arms completed the study but did not have histopathology results.
Measure: Count of Participants; unit: Participants
Groups:
- Mothers - 3 Dose SP: Women will be given SP (3 full strength tabs, 500 mg/25 mg) 3 times during pregnancy at 20, 28, and 36 weeks gestational age. In addition, placebos will be used to mimic the identical dosing strategy such that every 4 weeks women will receive two pills on day 1 (SP and placebo, DP and placebo, or two placebos) followed by one pill on days 2 and 3 (DP or placebo). Two placebos will be used, one that mimics the appearance of SP and one that mimics the appearance of DP.
  Infants will be given DP (once a day for 3 consecutive days using weight-based guidelines) every 12 weeks between 8 and 104 weeks of age. Infants randomized to receive DP every 12 weeks will receive placebo mimicking the dosing of DP every 4 weeks when they are not receiving study drug.
  3 dose sulfadoxine-pyrimethamine (SP) for adult women during pregnancy
  3-monthly dihydroartemisinin-piperaquine (DP) for infants
- Mothers - 3 Dose DP: Women will be given DP (3 full strength tabs, 40 mg/320 mg, given once a day for 3 consecutive days) 3 times during pregnancy at 20, 28, and 36 weeks gestational age. In addition, placebos will be used to mimic the identical dosing strategy such that every 4 weeks women will receive two pills on day 1 (SP and placebo, DP and placebo, or two placebos) followed by one pill on days 2 and 3 (DP or placebo). Two placebos will be used, one that mimics the appearance of SP and one that mimics the appearance of DP.
  Infants will be given DP (once a day for 3 consecutive days using weight-based guidelines) every 12 weeks between 8 and 104 weeks of age. Infants randomized to receive DP every 12 weeks will receive placebo mimicking the dosing of DP every 4 weeks when they are not receiving study drug.
  3 dose dihydroartemisinin-piperaquine (DP) for adult women during pregnancy
  3-monthly dihydroartemisinin-piperaquine (DP) for infants
- Mothers - Monthly DP: Women will be given DP (3 full strength tabs, 40 mg/320 mg, given once a day for 3 consecutive days) 3 times during pregnancy at 20, 28, and 36 weeks gestational age. In addition, placebos will be used to mimic the identical dosing strategy such that every 4 weeks women will receive two pills on day 1 (SP and placebo, DP and placebo, or two placebos) followed by one pill on days 2 and 3 (DP or placebo). Two placebos will be used, one that mimics the appearance of SP and one that mimics the appearance of DP.
  Infants will be given DP (once a day for 3 consecutive days using weight-based guidelines) every 4 weeks between 8 and 104 weeks of age.
  3 dose dihydroartemisinin-piperaquine (DP) for adult women during pregnancy
  Monthly dihydroartemisinin-piperaquine (DP) for infants
Arm/Group | Mothers - 3 Dose SP | Mothers - 3 Dose DP | Mothers - Monthly DP
Number analyzed (Participants) | 98 | 88 | 96
Participants | 49 | 30 | 26

2. Primary Outcome: Incidence of Malaria in Pregnant Women
Description: Incidence of malaria, defined as the number of incident episodes per time at risk. Incident cases will include all treatments for malaria not proceeded by another treatment in the previous 14 days.
Time Frame: Time at risk will begin after first dose of study drug and will end when study participants deliver or early study termination
Measure: Number; unit: events per person years
Arm/Group | Mothers - 3 Dose SP | Mothers - 3 Dose DP | Mothers - Monthly DP
Number analyzed (Participants) | 106 | 94 | 100
events per person years | 0.95 | 0.31 | 0

3. Primary Outcome: Incidence of Malaria in Infants
Description: Incident cases will include all treatments for malaria not proceeded by another treatment in the previous 14 days. The study investigators will test the hypotheses that A) infants born to mothers randomized to receive IPTp with 3 dose DP or monthly DP will have a lower incidence of malaria during the first 24 months of life compared to infants born to mothers who were randomized to receive IPTp with 3 doses of SP, and, B) infants randomized to receive monthly DP between 2-24 months of age will have a lower incidence of malaria between 24-36 months of age after the intervention is stopped compared to infants randomized q 3 monthly DP between 2-24 months of age.
Time Frame: Time at risk will begin at birth and will end when study participants reaches 24 months of age or early study termination (if prior to 24 months of age)
Population: All live births
Measure: Number; unit: Events per person years
Groups:
- 3 Dose SP Pregnancy / 3 Monthly DP Infancy: Women will be given SP (3 full strength tabs, 500 mg/25 mg) 3 times during pregnancy at 20, 28, and 36 weeks gestational age. In addition, placebos will be used to mimic the identical dosing strategy such that every 4 weeks women will receive two pills on day 1 (SP and placebo, DP and placebo, or two placebos) followed by one pill on days 2 and 3 (DP or placebo). Two placebos will be used, one that mimics the appearance of SP and one that mimics the appearance of DP.
  Infants will be given DP (once a day for 3 consecutive days using weight-based guidelines) every 12 weeks between 8 and 104 weeks of age. Infants randomized to receive DP every 12 weeks will receive placebo mimicking the dosing of DP every 4 weeks when they are not receiving study drug.
  3 dose sulfadoxine-pyrimethamine (SP) for adult women during pregnancy
  3-monthly dihydroartemisinin-piperaquine (DP) for infants
- 3 Dose DP Pregnancy / 3 Monthly DP Infancy: Women will be given DP (3 full strength tabs, 40 mg/320 mg, given once a day for 3 consecutive days) 3 times during pregnancy at 20, 28, and 36 weeks gestational age. In addition, placebos will be used to mimic the identical dosing strategy such that every 4 weeks women will receive two pills on day 1 (SP and placebo, DP and placebo, or two placebos) followed by one pill on days 2 and 3 (DP or placebo). Two placebos will be used, one that mimics the appearance of SP and one that mimics the appearance of DP.
  Infants will be given DP (once a day for 3 consecutive days using weight-based guidelines) every 12 weeks between 8 and 104 weeks of age. Infants randomized to receive DP every 12 weeks will receive placebo mimicking the dosing of DP every 4 weeks when they are not receiving study drug.
  3 dose dihydroartemisinin-piperaquine (DP) for adult women during pregnancy
  3-monthly dihydroartemisinin-piperaquine (DP) for infants
- 3 Dose DP Pregnancy / Monthly DP Infancy: Women will be given DP (3 full strength tabs, 40 mg/320 mg, given once a day for 3 consecutive days) 3 times during pregnancy at 20, 28, and 36 weeks gestational age. In addition, placebos will be used to mimic the identical dosing strategy such that every 4 weeks women will receive two pills on day 1 (SP and placebo, DP and placebo, or two placebos) followed by one pill on days 2 and 3 (DP or placebo). Two placebos will be used, one that mimics the appearance of SP and one that mimics the appearance of DP.
  Infants will be given DP (once a day for 3 consecutive days using weight-based guidelines) every 4 weeks between 8 and 104 weeks of age.
  3 dose dihydroartemisinin-piperaquine (DP) for adult women during pregnancy
  Monthly dihydroartemisinin-piperaquine (DP) for infants
- Monthly DP Pregnancy / 3 Monthly DP Infancy: Women will be given DP (3 full strength tabs, 40 mg/320 mg, given once a day for 3 consecutive days) every 4 weeks during pregnancy. In addition, placebos will be used to mimic the identical dosing strategy such that every 4 weeks women will receive two pills on day 1 (SP and placebo, DP and placebo, or two placebos) followed by one pill on days 2 and 3 (DP or placebo). Two placebos will be used, one that mimics the appearance of SP and one that mimics the appearance of DP.
  Infants will be given DP (once a day for 3 consecutive days) every 12 weeks between 8 and 104 weeks of age. Infants randomized to receive DP every 12 weeks will receive placebo mimicking the dosing of DP every 4 weeks when they are not receiving study drug.
  Monthly dihydroartemisinin-piperaquine (DP) for adult women during pregnancy
  3-monthly dihydroartemisinin-piperaquine (DP) for infants
- Monthly DP Pregnancy / Monthly DP Infancy: Women will be given DP (3 full strength tabs, 40 mg/320 mg, given once a day for 3 consecutive days) every 4 weeks during pregnancy. In addition, placebos will be used to mimic the identical dosing strategy such that every 4 weeks women will receive two pills on day 1 (SP and placebo, DP and placebo, or two placebos) followed by one pill on days 2 and 3 (DP or placebo). Two placebos will be used, one that mimics the appearance of SP and one that mimics the appearance of DP.
  Infants will be given DP (once a day for 3 consecutive days) every 4 weeks between 8 and 104 weeks of age.
  Monthly dihydroartemisinin-piperaquine (DP) for adult women during pregnancy
  Monthly dihydroartemisinin-piperaquine (DP) for infants
Arm/Group | 3 Dose SP Pregnancy / 3 Monthly DP Infancy | 3 Dose DP Pregnancy / 3 Monthly DP Infancy | 3 Dose DP Pregnancy / Monthly DP Infancy | Monthly DP Pregnancy / 3 Monthly DP Infancy | Monthly DP Pregnancy / Monthly DP Infancy
Number analyzed (Participants) | 101 | 44 | 49 | 48 | 52
Events per person years | 0.26 | 0.30 | 0.00 | 0.43 | 0.03

4. Primary Outcome: Incidence of Malaria in Infants
Description: as for outcome 3
Time Frame: Time at risk will begin at 24 months of age and will end when study participants reaches 36 months of age or termination
Population: All live births
Measure: Number; unit: Events per person years
Arm/Group | 3 Dose SP Pregnancy / 3 Monthly DP Infancy | 3 Dose DP Pregnancy / 3 Monthly DP Infancy | 3 Dose DP Pregnancy / Monthly DP Infancy | Monthly DP Pregnancy / 3 Monthly DP Infancy | Monthly DP Pregnancy / Monthly DP Infancy
Number analyzed (Participants) | 85 | 40 | 43 | 39 | 44
Events per person years | 0.87 | 0.88 | 0.83 | 1.24 | 0.64

5. Secondary Outcome: Number of Participants With Blood Samples Positive for Parasites by Microscopy or LAMP
Description: Prevalence of placental blood samples positive for parasites by microscopy or LAMP
Time Frame: Delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Mothers - 3 Dose SP | Mothers - 3 Dose DP | Mothers - Monthly DP
Number analyzed (Participants) | 96 | 88 | 96
Participants
  Micropscopic assessment of placental blood | 5 | 3 | 0
  LAMP assessment of placental blood | 19 | 3 | 2

6. Secondary Outcome: Number of Participants With Maternal Blood Samples Positive for Parasites by Microscopy and LAMP at Delivery
Description: Prevalence of maternal parasitemia at delivery by microscopy and LAMP
Time Frame: At delivery
Population: One observation in the monthly DP arm did not have results for microscopy; this outcome measure tests blood taken from the mother's arm (different from outcome measure 4 which tests blood taken from the placenta)
Measure: Number; unit: participants
Arm/Group | Mothers - 3 Dose SP | Mothers - 3 Dose DP | Mothers - Monthly DP
Number analyzed (Participants) | 102 | 89 | 98
participants
  Microscopy: number analyzed (Participants) | 102 | 89 | 97
  Microscopy | 5 | 1 | 0
  LAMP | 25 | 3 | 1

7. Secondary Outcome: Number of Participants With One or More Birth Outcomes: Congenital Malformations, Spontaneous Abortion, LBW (<2500g), Still Birth, Pre-term Delivery
Description: Congenital malformations, spontaneous abortion, LBW (<2500g), still birth, pre-term delivery
Time Frame: Delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Mothers - 3 Dose SP | Mothers - 3 Dose DP | Mothers - Monthly DP
Number analyzed (Participants) | 102 | 89 | 98
Participants | 19 | 19 | 9

8. Secondary Outcome: Prevalence of Anemia in Pregnant Women
Description: Prevalence of routine hemoglobin measurements < 11 g/dL
Time Frame: After first dose of study drugs up to delivery or early termination
Measure: Number; unit: hemoglobin measurements taken every 12wk
Units Other Than Participants: hemoglobin measurements taken every 12wk
Arm/Group | Mothers - 3 Dose SP | Mothers - 3 Dose DP | Mothers - Monthly DP
Number analyzed (Participants) | 106 | 94 | 100
Number analyzed (hemoglobin measurements taken every 12wk) | 269 | 237 | 258
hemoglobin measurements taken every 12wk | 94 | 72 | 61

9. Secondary Outcome: Incidence of Complicated Malaria in Infants
Description: Any treatment for malaria meeting criteria for severe malaria or danger signs
Time Frame: Birth up to 24 months of age or early study termination
Population: All live births
Measure: Number; unit: Events per person years
Arm/Group | 3 Dose SP Pregnancy / 3 Monthly DP Infancy | 3 Dose DP Pregnancy / 3 Monthly DP Infancy | 3 Dose DP Pregnancy / Monthly DP Infancy | Monthly DP Pregnancy / 3 Monthly DP Infancy | Monthly DP Pregnancy / Monthly DP Infancy
Number analyzed (Participants) | 101 | 44 | 49 | 48 | 52
Events per person years | 0.022 | 0.024 | 0.000 | 0.035 | 0.000

10. Secondary Outcome: Incidence of Hospital Admissions in Infants
Description: Admission to a hospital for pediatric inpatient care for any reason
Time Frame: Birth up to 24 months of age or early study termination
Measure: Number; unit: Events per person years
Arm/Group | 3 Dose SP Pregnancy / 3 Monthly DP Infancy | 3 Dose DP Pregnancy / 3 Monthly DP Infancy | 3 Dose DP Pregnancy / Monthly DP Infancy | Monthly DP Pregnancy / 3 Monthly DP Infancy | Monthly DP Pregnancy / Monthly DP Infancy
Number analyzed (Participants) | 101 | 44 | 49 | 48 | 52
Events per person years | 0.043 | 0.036 | 0.089 | 0.082 | 0.043

11. Secondary Outcome: Prevalence of Gametocytemia in Pregnant Women
Description: Proportion of urgent blood smears positive for gametocytes
Time Frame: Gestational age between 12-20 weeks (at study entry) up to delivery
Measure: Number; unit: Positive blood smears
Units Other Than Participants: Blood smears
Arm/Group | Mothers - 3 Dose SP | Mothers - 3 Dose DP | Mothers - Monthly DP
Number analyzed (Participants) | 106 | 94 | 100
Number analyzed (Blood smears) | 112 | 86 | 86
Positive blood smears | 4 | 1 | 3

12. Secondary Outcome: Prevalence of Parasitemia in Infants
Description: Proportion of routine monthly samples positive for parasites by LAMP. Proportion of routine samples (LAMP or blood smears) positive for asexual parasites.
Time Frame: Birth up to 24 months of age or early study termination
Measure: Number; unit: Positive blood smears
Units Other Than Participants: Blood smears
Arm/Group | 3 Dose SP Pregnancy / 3 Monthly DP Infancy | 3 Dose DP Pregnancy / 3 Monthly DP Infancy | 3 Dose DP Pregnancy / Monthly DP Infancy | Monthly DP Pregnancy / 3 Monthly DP Infancy | Monthly DP Pregnancy / Monthly DP Infancy
Number analyzed (Participants) | 101 | 44 | 49 | 48 | 52
Number analyzed (Blood smears) | 2378 | 1082 | 1155 | 1099 | 1208
Positive blood smears | 59 | 25 | 7 | 52 | 4

13. Secondary Outcome: Prevalence of Parasitemia at the Time of Monthly Routine Visits During Pregnancy
Description: Detection of malaria parasites by LAMP during pregnancy
Time Frame: After first dose of study drug through delivery or early termination
Measure: Number; unit: Positive specimens
Units Other Than Participants: Specimens
Arm/Group | Mothers - 3 Dose SP | Mothers - 3 Dose DP | Mothers - Monthly DP
Number analyzed (Participants) | 106 | 94 | 100
Number analyzed (Specimens) | 509 | 445 | 496
Positive specimens | 206 | 74 | 26

14. Secondary Outcome: Prevalence of Gametocytemia in Infants
Description: Proportion of routine blood smears positive for gametocytes
Time Frame: Birth up to 24 months of age or early study termination
Measure: Number; unit: Positive blood smears
Units Other Than Participants: Blood smears
Arm/Group | 3 Dose SP Pregnancy / 3 Monthly DP Infancy | 3 Dose DP Pregnancy / 3 Monthly DP Infancy | 3 Dose DP Pregnancy / Monthly DP Infancy | Monthly DP Pregnancy / 3 Monthly DP Infancy | Monthly DP Pregnancy / Monthly DP Infancy
Number analyzed (Participants) | 101 | 44 | 49 | 48 | 52
Number analyzed (Blood smears) | 2393 | 1087 | 1156 | 1102 | 1218
Positive blood smears | 7 | 1 | 0 | 4 | 0

ADVERSE EVENTS:
Time Frame: For women, from study drug initiation to 6 weeks postpartum or last observed date in study. For children, from study drug initiation to 4 weeks after last dose of study drugs.
Description: National Institutes of Health, Division of AIDS (DAIDS) Table for Grading the Severity of ADULT AND PEDIATRIC Adverse Events Version 1.0, December, 2004; clarification AUGUST 2009
Groups:
- Mothers - 3 Dose SP: Women were given SP (3 full strength tabs, 500 mg/25 mg) 3 times during pregnancy at 20, 28, and 36 weeks gestational age. In addition, DP placebo was used to mimic the identical dosing strategy such that every 4 weeks women will receive two pills on day 1 (SP and DP placebo) followed by one pill on days 2 and 3 (DP placebo).
- Mothers - 3 Dose DP: Women were given DP (3 full strength tabs, 40 mg/320 mg, given once a day for 3 consecutive days) 3 times during pregnancy at 20, 28, and 36 weeks gestational age. In addition, SP and DP placebos were used to mimic the identical dosing strategy as other arms such that every 4 weeks women will receive two pills on day 1 (DP and SP placebo) followed by one pill on days 2 and 3 (DP placebo).
- Mothers - Monthly DP: Women were given DP (3 full strength tabs, 40 mg/320 mg, given once a day for 3 consecutive days) monthly. In addition, SP placebo to mimic the identical dosing strategy as other arms such that every 4 weeks women will receive two pills on day 1 (DP and SP placebo) followed by one pill on days 2 and 3 (DP).
- Infants - Monthly DP: DP half-strength tablets given once a day for 3 consecutive days according to weight based guidelines.
- Infants - 3 Monthly DP: DP half-strength tablets given once a day for 3 consecutive days according to weight based guidelines. Infants received placebo mimicking the dosing of DP every 4 weeks when they are not receiving study drug.
Arm/Group | Mothers - 3 Dose SP | Mothers - 3 Dose DP | Mothers - Monthly DP | Infants - Monthly DP | Infants - 3 Monthly DP
All-Cause Mortality (participants affected / at risk) | 0/106 | 0/94 | 0/100 | 4/100 | 3/191
Serious Adverse Events (participants affected / at risk) | 6/106 | 9/94 | 3/100 | 9/100 | 15/191
Other Adverse Events (participants affected / at risk) | 90/106 | 78/94 | 89/100 | 94/100 | 183/191
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mothers - 3 Dose SP (N=106) | Mothers - 3 Dose DP (N=94) | Mothers - Monthly DP (N=100) | Infants - Monthly DP (N=100) | Infants - 3 Monthly DP (N=191)
Anemia (Blood and lymphatic system disorders) | 2 (2) | 1 (1) | 2 (2) | 3 (3) | 1 (1)
Congenital Anomaly (Congenital, familial and genetic disorders) | 2 (2) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Stillbirth (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Threatened Abortion (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Retained products of conception (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Preeclampsia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyelonephritis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 3 (3)
Elevated temperature (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Elevated Alanine Aminotransferase (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Intestinal Obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Altered Mental State (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Burns (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neutropenia (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Malnutrition (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dehydration (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mothers - 3 Dose SP (N=106) | Mothers - 3 Dose DP (N=94) | Mothers - Monthly DP (N=100) | Infants - Monthly DP (N=100) | Infants - 3 Monthly DP (N=191)
Abdominal pain (General disorders) | 74 (172) | 58 (122) | 73 (132) | 0 (0) | 0 (0)
Cough (General disorders) | 55 (94) | 48 (71) | 57 (77) | 94 (1127) | 183 (2230)
Headache (General disorders) | 56 (90) | 45 (70) | 55 (78) | 0 (0) | 0 (0)
Chills (General disorders) | 20 (21) | 13 (14) | 11 (12) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 10 (12) | 8 (10) | 10 (13) | 87 (470) | 168 (938)
Malaise (General disorders) | 15 (16) | 9 (9) | 6 (8) | 10 (10) | 25 (28)
Dysphagia (General disorders) | 9 (9) | 2 (2) | 13 (14) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 7 (8) | 8 (8) | 8 (8) | 58 (114) | 117 (191)
Nausea (Gastrointestinal disorders) | 2 (2) | 4 (4) | 2 (2) | 0 (0) | 0 (0)
Urinary tract infection (Renal and urinary disorders) | 3 (3) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Anorexia (General disorders) | 2 (2) | 0 (0) | 4 (4) | 16 (18) | 43 (191)
Anemia (Blood and lymphatic system disorders) | 9 (10) | 2 (3) | 4 (4) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 29 (43) | 56 (191)
Conjunctivitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 27 (34) | 49 (62)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-10-25): https://cdn.clinicaltrials.gov/large-docs/47/NCT02163447/Prot_001.pdf
  • Statistical Analysis Plan (2015-05-08): https://cdn.clinicaltrials.gov/large-docs/47/NCT02163447/SAP_000.pdf